CLINICAL TRIAL: NCT00942695
Title: Energy Value of Macronutrients From Pistachio Nuts and Mechanisms of Nutrient Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Collaborators: Paramount Farms (Unknown)
Responsible Party: David J. Baer, Ph. D., Principal Investigator, USDA-ARS
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2009-109
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Energy; Cardiovascular Disease; Cancer
Keywords: pistachio; nuts; energy value; cardiovascular disease; phytonutrient; gene expression; energy value of pistachio nuts
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- base (Other): average American diet without pistachios
  Interventions: Other: control
- 1.5PD (Active Comparator): average American diet plus 1.5 oz per day pistachios
  Interventions: Other: 1.5PD
- 3.0PD (Active Comparator): average American diet plus 3.0 oz per day pistachios
  Interventions: Other: 3.0PD

INTERVENTIONS:
Other: 1.5PD — average American diet plus 1.5 oz per day pistachios
  Arms: 1.5PD
Other: 3.0PD — average American diet plus 3.0 oz per day pistachios
  Arms: 3.0PD
Other: control — average American diet without pistachios
  Arms: base

SUMMARY:
The objective of this study is to measure the energy value of pistachios in the human diet and study molecular mechanisms that may help explain the beneficial health effects of pistachios.

DETAILED DESCRIPTION:
Previous studies have suggested that nut consumption imparts a variety of health benefits, including reduction of cardiovascular disease and improved satiety. However, studies of pistachios are extremely limited. The aim of this study is to determine the energy value of pistachios in the human diet and to probe mechanisms by which pistachios impart health benefits. The metabolizable energy value of pistachio nuts will be calculated based on the chemical composition and energy content of the consumed diet and excreta. This will provide a better estimate of the energy value of pistachios than simply calculating energy value based on Atwater factors. In addition to determining the energy value of pistachios, we will evaluate the effects of pistachio-rich diets on plasma phytonutrient levels and on gene expression changes to determine what protective mechanisms are activated by pistachio consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 65 years at beginning of study
* BMI between 20 and 38 kg/m2
* Fasting glucose < 126 mg/dl
* Blood pressure < 160/100 (controlled with certain medications)
* Fasting total blood cholesterol < 280 mg/dl
* Fasting triglycerides < 300 mg/dl

Exclusion Criteria:

* Presence of kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of bariatric or certain other surgeries related to weight control
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* Antibiotic use during the intervention or for 3 weeks prior to any intervention period
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 12 months or who plan to initiate a weight loss program during the next 10 months
* Known (self-reported) allergy or adverse reaction to pistachios or other nuts
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
to measure the energy value of pistachios in the human diet | 3 weeks

SECONDARY OUTCOMES:
to study molecular mechanisms that may help explain the beneficial health effects of pistachios | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David J Baer, Ph. D., Principal Investigator — United States Department of Agriculture (USDA)
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States